CLINICAL TRIAL: NCT01727739
Title: Tibial Tunnel Widening in ACL Reconstruction-Comparing Two Bioscrews: A Prospective Randomized Clinical Trial
Brief Title: Tibial Tunnel Widening in Anterior Cruciate Ligament (ACL) Reconstruction-Comparing Two Bioscrews
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Responsible Party: Principal Investigator, Peter MacDonald, Research Associate, Panam Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2012:059
Record Dates: First submitted 2012-11-07; First posted 2012-11-16 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: ACL
Keywords: Tibial tunnel widening; Interference screws

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- PLLA bioscrew (Active Comparator): poly-L-lactic acid bioscrew
  Interventions: Device: Linvatec PLLA
- PLLA+TCP bioscrew (Active Comparator): poly-l-lactic acid with beta tricalcium phosphate bioscrew
  Interventions: Device: Linvatec PLLA+TCP

INTERVENTIONS:
Device: Linvatec PLLA+TCP — Linvatec PLLA+TCP tibial interference screw fixation will be used in ACL reconstruction.
  Arms: PLLA+TCP bioscrew
Device: Linvatec PLLA — Linvatec PLLA tibial interference screw fixation will be used in ACL reconstruction.
  Arms: PLLA bioscrew

SUMMARY:
Widening of the single tibial tunnel following ACL surgery with quadrupled hamstrings autograft may contribute to failure of the graft and/or present technical challenges secondary to bone loss in a revision setting (Getelman, 1999). As such, efforts should be made to minimize the incidence and magnitude of tibial tunnel widening without sacrificing the biomechanical properties of the graft construct. The purpose of this investigation is to examine the tibial tunnel widening relationship between bioabsorbable interference screws composed of poly-L-lactic acid (PLLA) alone and composite bioabsorbable interference screws composed of poly-L-lactic acid embedded with beta tricalcium phosphate (PLLA+TCP) utilized as tibial fixation devices.

Specifically the study has the following objectives: 1) To quantify the extent of tibial tunnel enlargement at 3-, 6- and 12-months post ACL reconstruction with autogenous quadrupled hamstring graft; 2) To determine if the incorporation of beta tricalcium phosphate to the bioabsorbable interference screw alters the observed magnitude of tunnel widening; 3) To hypothesize mechanisms for any observed differences between tibial fixation devices; and 4) To correlate tibial tunnel widening with clinical outcome status. It is hypothesized that the PLLA+TCP bioabsorbable interference screw will not be associated with a reduction in tibial tunnel widening around the implant but rather between the implant and articular surface, compared to the PLLA alone screw. It is also hypothesized that there will be no effect of observed tunnel widening on clinical outcomes or graft failure rates.

ELIGIBILITY:
Inclusion Criteria:

* Must have a unilateral ACL rupture
* Patients must be between 18 and 45 years old

Exclusion Criteria:

* Concomitant medial collateral, lateral collateral, or posterior collateral ligament tears
* Severe chondromalacia or severe meniscal tear
* Previous history of ipsilateral knee joint pathology, surgery, or trauma to that knee
* Unwillingness to be followed for 12 months post-operatively
* History of arthritis (osteoarthritis or rheumatoid)
* Pregnancy
* Psychiatric illness that precludes informed consent
* Unable to speak or read English/French
* Major medical illness (life expectancy less than 1 year or unacceptably high operative risk)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Radiographs | 12 months post op
  At 3-, 6- and 12-months post-operatively, subjects will undergo radiographic examination of their affected knee (standardized AP and lateral views) for analysis of tibial tunnel parameters. Radiographic analysis will be conducted by a single orthopaedic surgeon/fellow/resident blinded to subject group and clinical examination results. Parameters to be recorded and analyzed according to a standardized method: tibial tunnel diameter (max/min).
  We will also look for: Evidence of lysis in the tunnel and changes in morphological features of tunnel over time

SECONDARY OUTCOMES:
ACL Quality of Life Scores | 12 months post op
  Completed at 3-, 6- and 12-months post operatively for subjective outcome measure.

OTHER OUTCOMES:
IKDC Assessment | 12 months post op
  Range of motion assessment at 3-,6-and 12-months post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Peter B MacDonald, MD FRCS(C), Principal Investigator — Pan Am Clinic
Locations (1):
- Pan Am Clinic, Winnipeg, Manitoba, Canada